CLINICAL TRIAL: NCT05145153
Title: Incidence of Chronic Pain After Thoracic Surgery
Status: Recruiting | Type: Observational
Sponsor: Atatürk Chest Diseases and Chest Surgery Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Musa Zengin, Principal İnvestigator, Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Other Study IDs: 2012-KAEK-15/2378
Record Dates: First submitted 2021-11-18; First posted 2021-12-06 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-05

CONDITIONS: Postoperative Pain; Postoperative Pain, Acute; Postoperative Pain, Chronic; Video-Assisted Thoracoscopic Surgery; Thoracotomy
Keywords: Postoperative Pain; Postoperative Pain, Acute; Postoperative Pain, Chronic; Video-Assisted Thoracoscopic Surgery; Thoracotomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Thoracic surgery application — The chronic pain findings of the patients who underwent thoracic surgery will be questioned at the postoperative 3rd and 6th months.

SUMMARY:
Thoracotomy and video-assisted thoracic surgery procedures are frequently performed in thoracic surgery. It is widely accepted that thoracotomy causes severe acute pain. This prolongs the discharge time of the patients, and increases the frequency of postoperative pulmonary complications and postoperative morbidity. Postoperative acute pain may cause chronic thoracotomy pain in the later period, and may adversely affect the quality of life of the patients. Video-assisted thoracic surgery (VATS) has become the standard procedure in minor and major lung surgeries. Postoperative pain is seen in patients undergoing VATS, although it is not as severe as after thoracotomy. As in thoracotomy, this affects the postoperative pulmonary complications and the discharge time of the patients. Likewise, this pain can cause chronic pain.

In this study, it was aimed to analyze the symptoms of chronic pain in the 3rd and 6th months postoperatively in patients who had undergone thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* American Society of Anesthesiologists physical status I-II-III
* Body mass index between 18-35 kg/m2
* Patients undergoing elective thoracic surgery

Exclusion Criteria:

* Advanced cancer
* History of chronic analgesic therapy
* Patients with previous thoracic surgery
* Patients who were operated under emergency conditions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18-65 years, in the ASA I-II-III risk group, with a BMI between 18-35 kg/m2 and undergoing thoracic surgery will be included in our study.
  Patients under the age of 18 years and over the age of 65 years, with an ASA score of IV and above, with a BMI below 18 kg/m2 and above 35 kg/m2, who were operated under emergency conditions, and who received chronic pain treatment will be excluded from the study.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-10-08 (Estimated); Study Completion 2024-11-28 (Estimated)

PRIMARY OUTCOMES:
Pain scores at 3th months. | Chronic pain symptoms at 3th months.
  Choronic pain symptoms will be assessed using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Neuropathic pain symptoms (Burning, stabbing, electric shock-like pain, tingling, numbness, pins and needles feeling, hyperalgesia, allodynia, and hypoesthesia) will also be asked to the patients in the 3rd month after surgery.
Pain scores at 6th months. | Chronic pain symptoms at 6th months.
  Choronic pain symptoms will be assessed using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain). Neuropathic pain symptoms (Burning, stabbing, electric shock-like pain, tingling, numbness, pins and needles feeling, hyperalgesia, allodynia, and hypoesthesia) will also be asked to the patients in the 6th month after surgery.

SECONDARY OUTCOMES:
Life quality | The effect of chronic pain on quality of life at 3rd and 6th months.
  It will be questioned whether chronic pain affects the patient's quality of life.
  1. has no affect
  2. has little effect
  3. has medium affect
  4. has a lot of affects

CONTACTS AND LOCATIONS:
Overall Officials: Musa Zengin, MD, Principal Investigator — Atatürk Chest Diseases and Chest Surgery Training and Research Hospital
Locations (1):
- Ankara Atatürk Chest Disease and Chest Surgery Training and Research Hospital, Keçiören, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No